CLINICAL TRIAL: NCT03254095
Title: Thermal and Biomechanical Characterization of Diabetic Foot Patients, Predictors of Skin Temperature, Barefoot Plantar Pressure and Ulceration.
Brief Title: Predictors of Skin Temperature, Plantar Pressure and Ulceration in Diabetic Foot Patients.
Status: Completed | Type: Observational
Sponsor: Universidade do Porto (Other)
Collaborators: Centro Hospitalar do Porto (Other)
Responsible Party: Principal Investigator, Adérito Seixas, PhD Student, Universidade do Porto
Other Study IDs: FADEUP_PhD_AdéritoSeixas#1
Record Dates: First submitted 2017-08-12; First posted 2017-08-18 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Diabetic Foot; Diabetes
Keywords: Skin temperature; Plantar pressure; Diabetic foot; Tissue hardness; Neuropathy; Peripheral artery disease
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

SUMMARY:
Diabetes is a chronic disease with increasing prevalence worldwide with a high burden to individuals and the society and it is expected to be the 7th leading cause of death in 2030. Diabetes related complications manifest in many body parts, often in the foot, due to reduced blood flow and nerve damage, increasing the risk of ulcers and amputation. High plantar pressures during walking contribute to the development of foot ulcers and foot ulcer recurrence. Emerging studies also point skin temperature as another predictor of foot ulceration. However, the number of studies including prediction models of plantar pressure and skin temperature are scarce, especially in patients with confirmed diagnosis of diabetic foot and a history of foot ulcer. Factors like mobility, hardness of plantar soft tissue, foot deformities and other diabetes related characteristics have been related to plantar pressure measurements but not to foot skin temperature measurements, and the relation between skin temperature and plantar pressure has not been much explored in the literature. The role of these variables in the development of foot ulceration needs further attention, especially in patients with history of foot ulcers has they are at the highest risk to develop a foot ulcer.

Therefore, the goal of this research is to determine which variables can be used to predict plantar pressure and skin temperature and which factors are associated with the development of foot ulcers in patients with established diagnosis of diabetic foot. The associations between skin temperature and plantar pressure will also be addressed.

ELIGIBILITY:
Inclusion Criteria:

* Adults (over 18 years)
* Diagnosed as diabetic foot patient
* Able to walk 10 meters without assistance

Exclusion Criteria:

* Non-cooperating patients
* Patients with major amputations
* Patients with a draining ulcer and/or infection
* Patients with cognitive impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with established diagnosis of diabetic foot. Diabetic Foot is related to infection, ulceration or destruction of tissues of the foot associated with neuropathy and/or peripheral artery disease in the lower extremity of people with diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Skin temperature | At study entry
  After an acclimation period of 10 minutes, skin temperature of the sole and dorsum of the foot will be assessed with a thermographic camera. Thermograms will be captured before, immediately after and five minutes after a two-minute cold stress test using an aluminium plaque.
Barefoot plantar pressure | At study entry
  Barefoot plantar pressure will be assessed using a pressure platform.
Percentage of patients developing a foot ulcer | One year after enrollment
  The occurrence of foot ulceration will be assessed during a period of 1 year.

SECONDARY OUTCOMES:
Ankle mobility | At study entry
  Active ankle mobility (dorsiflexion and plantarflexion) will be assessed with a goniometer.
Hallux active extension range of movement | At study entry
  Hallux active extension mobility will be assessed with a goniometer.
Soft tissue hardness | At study entry
  Soft tissue hardness will be assessed with a durometer.
In-shoe plantar pressure | At study entry
  In-shoe plantar pressure will be assessed using an insole system.
Time to ulceration | At study entry
  The time to ulcer occurrence will be assessed.

OTHER OUTCOMES:
Disease duration | At study entry
  Diabetes duration until the assessment day will be noted.
Type of diabetes | At study entry
  The type of diabetes (Type I or Type II) will be assessed.
Foot deformity | At study entry
  The presence of claw toes, hammer toes, hallux valgus, flat foot, increased foot arch and Charcot will be assessed.
Amputation | At study entry
  The presence of minor amputation will be assessed.
Neuropathy | At study entry
  The presence of neuropathy will be assessed according to the criteria of the International Working Group on the Diabetic Foot.
Peripheral artery disease | At study entry
  Peripheral artery disease signs - an absence of foot pulses and intermittent claudication - will be assessed.
Generic health status | At study entry
  The generic health status will be assessed with the EQ-5D-5L instrument.
Age | At study entry
  The age of participants at the assessment day will be noted.
Height | At study entry
  The height of participants at the assessment day will be noted.
Weight | At study entry
  The weight of participants at the assessment day will be noted.
Body mass index | At study entry
  Body mass index will be calculated from the height and weight of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Adérito RD Seixas, MSc, Principal Investigator — Universidade do Porto